CLINICAL TRIAL: NCT06191029
Title: Translation and Validation of Cognitive Failure Questionniare in Urdu Among Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIUaniqa
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Elderly Population

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults
  Interventions: Behavioral: Urdu translated cognitive failure questionnaire

INTERVENTIONS:
Behavioral: Urdu translated cognitive failure questionnaire — Urdu Translated version of cognitive failure questionnaire will be given to adults to fill it accordingly and then it's reliability and validity will be checked

SUMMARY:
study is based on translation of Cognitive Failure questionnaire in URDU and thrn to check its reliability an Validation in Elderly

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients Participants belonging to Urdu speaking class.

Age should above 60 years Participants should be capable to complete the questionnaire without any help. Participants with mild cognitive impairment.

Exclusion Criteria:

* Individual below 60 years. Participants not capable to complete the questionnaire without any help. Participant who can't understand urdu

Ages: 55 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the adult's having age above 60 years and able to read Urdu by themselves
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Translation and validity of cognitive failure questionnaire in Urdu | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Aniqa Khalid, MsNmpt, Principal Investigator — Riphah
Locations (1):
- Aniqa, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No